CLINICAL TRIAL: NCT00523120
Title: Topical Voltaren as an Alternative Treatment for Otitis Externa
Brief Title: Topical Voltaren in Otitis Externa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sieff Medical Center (Other)
Responsible Party: Principal Investigator, victor kizhner, Victor Kizhner MD, Sieff Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP 7-264S
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Otitis Externa
MeSH Terms: conditions — Otitis Externa | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): voltaren ophta
  Interventions: Drug: diclofenac sodium
- 2 (Active Comparator): dexotic
  Interventions: Drug: dexotc

INTERVENTIONS:
Drug: diclofenac sodium — topical solution used in ear 5 drops 8 3/day
  Other Names: voltaren ophta
  Arms: 1
Drug: dexotc — aural drops
  Other Names: dexotic
  Arms: 2

SUMMARY:
Voltaren being a Non-steroidal anti-inflammatory drug (NSAID) drug may be used as a single drug therapy in otitis externa being both therapeutic and analgesic thus reducing consumption of oral analgesia.

DETAILED DESCRIPTION:
anticipated advantages are: reduction of inflammation and edema, no fungal overpopulation- when steroids are employed, contains boric acid as an ingredient, high safety profile, can be switched to antibiotic therapy later, can be used in conjunction wit steroids

ELIGIBILITY:
Inclusion Criteria:

* Adults having otitis externa as single diagnosis mild to moderate

Exclusion Criteria:

* Diabetes
* Children
* Pregnant women
* Immune compromise
* Starting other treatment
* Moderate to severe otitis externa

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
reducing oral analagestic use | 1 week

SECONDARY OUTCOMES:
adding an alternative treatment for otitis externa | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: victor kizhner, m.d., Principal Investigator — Sieff Medical Center, Safed, ISRAEL
Locations (1):
- Sieff Medical Center, Safed, Israel

REFERENCES:
- See also: Sieff Medical Center — http://www.ziv.org.il/